CLINICAL TRIAL: NCT05494996
Title: Psychometric Properties of the Chinese Version of the Five-item Relationship Satisfaction Scale
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, Associate Professor, Sun Yat-sen University
Other Study IDs: wjn-RS5
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Relationship, Family
Keywords: Factor Analysis, Statistical; Psychometrics / methods; Family Relations / psychology*

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaires assessed partners: 1. ≥18 years old;
  2. Participants who are married or in a romantic relationship;
  3. Be able to read and communicate in Chinese.
  Interventions: Other: Questionnaires set

INTERVENTIONS:
Other: Questionnaires set — Participants will be asked to respond to the demographic information sheet and the five-item relationship satisfaction scale(RS5) .

SUMMARY:
The aims of this study are to translate the five-item relationship satisfaction scale（RS5) into Chinese and assess its psychometric properties among Chinese patients.

DETAILED DESCRIPTION:
This study will use forward translation, reverse translation, and comprehensive methods to translate the RS5 scale into Chinese ,which will be more in line with the Chinese language and cultural environment. This study will also verify its reliability and validity in a large sample population to form a formal version of the scale. The scale will provide an effective tool for evaluating the degree of relationship satisfaction in China.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old;
* Participants who are married or in a romantic relationship;
* Be able to read and communicate in Chinese.

Exclusion Criteria:

* Those who are unable to communicate due to serious mental or physical illnesses such as deafness, confusion caused by mental illness, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total number of 278 spouses/partners who are married or in a romantic relationship.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Relationship satisfaction | Baseline
  The five-item relationship satisfaction scale（RS5）is a validated self-reported instrument assessing e-cigarette dependence.It consists of five items which are rated on a 6-point Likert scale (1 = Strongly disagree, 6 = Strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- XIAW, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The non-identified individual participant data will be shared after the outcomes have been published.
Supporting Information: SAP
Time Frame: After the publication of the study
Access Criteria: Researchers should contact the PI for approval of the study protocol.